CLINICAL TRIAL: NCT05769959
Title: An Open-Label, Multicenter, Phase 1 Study to Evaluate Safety, Pharmacokinetics, and Preliminary Anti-Tumor Activity of RO7515629 in Participants With Unresectable and/or Metastatic HLA-G Positive Solid Tumors
Brief Title: Study of RO7515629 in Participants With HLA-G Positive Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision (not related to safety, efficacy or quality).
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BP44068
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Renal Cell Carcinoma; Non-small Cell Lung Cancer; Pancreatic Adenocarcinoma; Colorectal Cancer; Ovarian Neoplasms
Keywords: HLA-G; Human leukocyte antigen G; Renal cell carcinoma; Non-small cell lung cancer; Pancreatic adenocarcinoma; Colorectal cancer; Epithelial ovarian cancer; Primary peritoneal cancer; Fallopian tube cancer; RO7515629; Tocilizumab
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part I Single Participant Cohort RO7515629 Dose Escalation (Experimental): Participants will receive a fixed dose of RO7515629 intravenously as a single agent on cycle 0 day -7 and 7 days later on cycle 1 day 1 followed by every three-week dosing frequency. Treatment may continue for up to 12 months maximum or until progression, loss of clinical benefit, intolerable toxicity, withdrawal from study treatment or death.
  Interventions: Drug: RO7515629; Drug: tocilizumab
- Part II Multiple Participant Cohort RO7515629 Dose Escalation (Experimental): Participants will receive RO7515629 intravenously, as a single agent on cycle 0 day -7 and 7 days later on cycle 1 day 1 followed by every three-week dosing frequency. In case of toxicity, step up dosing (single or double) may be implemented. Treatment may continue for up to 12 months maximum or until progression, loss of clinical benefit, intolerable toxicity, withdrawal from study treatment or death.
  Interventions: Drug: RO7515629; Drug: tocilizumab
- Part III Multiple Participant Cohort RO7515629 Dose Expansion (Experimental): Participants with selected solid tumors will receive a selected dose of RO7515629 intravenously as a single agent based on the recommended dose sequence for expansion (RDE) and dosing regimen selected from Part I and Part II. Treatment may continue for up to 12 months maximum or until progression, loss of clinical benefit, intolerable toxicity, withdrawal from study treatment or death.
  Interventions: Drug: RO7515629; Drug: tocilizumab

INTERVENTIONS:
Drug: RO7515629 — RO7515629 will be administered intravenously at a dose and schedule as specified for the respective study part and cohort.
Drug: tocilizumab — Tocilizumab will be used as rescue medication only. Tocilizumab will be administered as required for the management of cytokine release syndrome (CRS).
  Other Names: Actemra, RoActemra

SUMMARY:
The main purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, immune response and preliminary anti-tumor activity of RO7515629 alone in participants with advanced or metastatic solid tumors expressing human leukocyte antigen G (HLA-G).

ELIGIBILITY:
Inclusion Criteria:

* Unresectable and/or metastatic HLA-G-positive solid tumors, for which standard therapy does not exist, or has proven to be ineffective or intolerable
* Confirmed HLA-G tumor expression.
* Radiologically measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Life expectancy of at least 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematological, liver, renal and pulmonary function
* Willingness to abide by protocol defined contraceptive requirements for the duration of the study.

Exclusion Criteria:

* History or clinical evidence of Central Nervous System (CNS) metastases unless protocol specified criteria are met
* Leptomeningeal metastases
* Rapid disease progression including lesions that are a threat to vital organs or non-irradiated lesions 2cm or larger at critical sites where tumor swelling may pose a risk to critical anatomical structures
* Participants with another invasive malignancy in the last 2 years unless protocol specified criteria are met
* Uncontrolled hypertension
* Active interstitial lung disease (ILD), pneumonitis or a history of ILD/pneumonitis requiring treatment with steroids, history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest Computed Tomography (CT) scan
* Participants with central cavitation or tumor(s) shown to be invading or abutting major blood vessels by imaging or the Investigator determines the tumor(s) is likely to invade major blood vessels and cause fatal bleeding
* Participants with pulmonary military metastatic pattern or pulmonary lymphangitic carcinomatosis
* History of pulmonary embolism within 3 months prior to study entry
* Significant cardiovascular disease
* Presence of active or uncontrolled infection or any major episode of infection requiring treatment with IV antibiotics or hospitalization within 4 weeks prior to initiation of study treatment.
* Known hepatitis B or C (actively replicating) based on protocol specified criteria
* Known Human Immunodeficiency Virus (HIV) positivity
* Presence of an indwelling line or drain
* Active auto-immune disease that has required systemic therapy within the past 2 years unless protocol specified exceptions are met
* Major surgery within 28 days prior to first study treatment
* Last treatment with anti-cancer therapy or any investigational drug 28 days or less prior to the first study treatment
* Last dose of immunostimulating or immunosuppressive therapy 28 days or less prior to the first study treatment
* Regular dose of corticosteroids that exceeds prednisone 10 mg/day or equivalent within 28 days prior to first study treatment
* Prior treatment with T cell engaging or adoptive cell therapy
* Administration of a live, attenuated vaccine 28 days or less prior to first study treatment
* Contraindication or known hypersensitivity to any of the components of RO7515629 or tocilizumab or dexamethasone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Part 1, 2, 3: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 15 months
Part 1 and 2: Number of Participants With Dose Limiting Toxicities (DLTs) | From start of study treatment (cycle 0 day -7 or cycle 0 day -14) until two weeks after second or third RO7515629 infusion (cycle 1 day 1) for a total DLT window of up to 28 days.

SECONDARY OUTCOMES:
Part 1, 2, 3: Pharmacokinetic Analysis: Maximum Serum Concentration (Cmax) of RO7515629 | Up to 13 months
Part 1, 2, 3: Pharmacokinetic Analysis: Time of Maximum Serum Concentration (Tmax) of RO7515629 | Up to 13 months
Part 1, 2, 3: Pharmacokinetic Analysis: Minimum Serum Concentration (Cmin) of RO7515629 | Up to 13 months
Parts 1, 2, 3: Pharmacokinetic Analysis: Clearance (CL) of RO7515629 | Up to 13 months
Part 1, 2, 3: Pharmacokinetic Analysis: Volume of Distribution at Steady State (Vss) of RO7515629 | Up to 13 months
Part 1, 2, 3: Pharmacokinetic Analysis: Area Under The Curve (AUC) of RO7515629 | Up to 13 months
Part 1, 2, 3: Number of Participants With RO7515629 Anti-drug Antibodies (ADAs) | Up to 13 months
Part 1, 2, 3: Objective Response Rate (ORR) | Up to approximately 18 months
Part 1, 2, 3: Disease Control Rate (DCR) | Up to approximately 18 months
Part 1, 2, 3: Duration of Response (DoR) | Up to approximately 18 months
Part 1, 2, 3: Progression Free Survival (PFS) | Up to approximately 18 months
Part 1, 2, 3: Overall survival (OS) | Up to approximately 18 months
  Defined as the time from first dose of study treatment to time of death.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- United States (2):
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - SCRI Oncology Partners, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No